CLINICAL TRIAL: NCT00912834
Title: Urine Analysis in Different Types of Athletes
Brief Title: Study of Prevalence of Proteinuria, Urinary Tract Infection or Hematuria in Athletes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: FarEasternMH, hospital
Other Study IDs: 97088
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-06

CONDITIONS: Proteinuria
Keywords: hematuria; urinary tract infection
MeSH Terms: conditions — Proteinuria; Hematuria; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 1: tract and field athletes
- 2: swimming athletes
- 3: tennis athletes
- 4: football athletes
- 5: basketball athletes
- 6: Badminton athletes
- 7: control group

SUMMARY:
To understand the urine analysis of athletes

DETAILED DESCRIPTION:
there maybe some genitourinary problem related to athletes, such as proteinuria, hematuria, scrotal pain, STD, etc. To explore these problems and give adequate management for them not only improved athletes' health, but also it can do their best in their exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* proteinuria, hematuria, pyuria

Exclusion Criteria:

* bacteriuria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In some types exercise, including basketball, swimming, tract & field, tennis, football athletes, we make a study analysis of their urine data to find any abnormality such as microhematuria, proteinuria or pyuria.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Estimated); Study Completion 2009-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yin Wu, MD, Study Chair — Chung Yin Wu